CLINICAL TRIAL: NCT01372696
Title: A Correlation of the Endoscopic Characteristics of Colonic LSTs With Their Somatic or Germline Mutations. A Prospective, Genome Wide Study
Brief Title: Endoscopic Characteristics of Colonic Tumours
Acronym: C-LST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study abandoned
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Dr Michael Bourke, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LST-SGM
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyp; Colon Cancer
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue sample (Other): Patients who consent to participate in this study will have a small sample of their polyp and normal tissue sent for molecular testing.
  Interventions: Other: Sample of polyp

INTERVENTIONS:
Other: Sample of polyp — A small sample of the colonic polyp will be obtained for molecular testing. The remaining polyp will be sent for regular histological testing

SUMMARY:
The purpose is to investigate whether polyps that look different at colonoscopy, have formed via different mutations and have different risks of turning into cancer.

DETAILED DESCRIPTION:
Laterally spreading tumours (LSTs), are polyps that have a lateral extension along the colon wall with minimal vertical growth. It has become evident over the last few years that rather than being a single entity requiring an accumulation of mutations, colon cancer is in fact a heterogenous disease forming via multiple distinct genetic pathways. Additionally, with improved endoscopic characterization, it has been noted from experience at Westmead hospital that two macroscopically distinct types of LSTs, "granular" and "non granular", have different natural histories and risks of invasive cancer. It is therefore hypothesised that different polyp types have different genetic abnormalities, and potentially form via distinct genetic pathways, although this theory has not been widely examined.

This knowledge would be important in furthering our understanding of the development of cancer. There is accumulating evidence that genetic abnormalities may be a better predictor of cancer behaviour than histological grade. Additionally, guidelines for colonoscopy surveillance are currently a one size fits all approach that do not reflect the genetic heterogeneity of the disease and the knowledge that only 5% of polyps progress to cancer. Genetic studies may assess future cancer risk to a person in polyps once removed and plan surveillance colonoscopy frequency. This is an area with interest currently due to the national bowel cancer screening programme, with obvious cost implications for decision makers.

ELIGIBILITY:
Inclusion Criteria:

* Intention to perform Endoscopic Mucosal Resection
* Polyp equal to or greater than 20mm
* over 18 years of age
* Able to give informed consent to involvement in trial

Exclusion Criteria:

* Pregnancy
* Lactation: currently breastfeeding
* Taken clopidogrel within 7 days
* Taken warfarin within 5 days
* Had full therapeutic dose unfractionated heparin within 6 hours
* Had full therapeutic dose low molecular weight heparin (LMWH) within 12 hours
* Known clotting disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Significant differences in molecular abnormalities. | Samples will be looked at and stored for approx 15 years
  The aim of this project is to look for statistically significant differences in molecular abnormalities from the three known genetic pathways, between the two different morphological types, granular and non-granular, to potentially demonstrate that these different polyps form via different genetic pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, Principal Investigator — Westmead Hospital - Endoscopy Unit
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia